CLINICAL TRIAL: NCT04088344
Title: The Relative Contribution of Dietary Lipids vs. of Fatty Acids to Non-adipose Tissues and the Effect of a Carbohydrate-rich Diet in Healthy Subjects
Brief Title: Effect of a Carbohydrate-rich Diet in Healthy Subjects
Acronym: AGL9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, André Carpentier, tenured professor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: 2013-530, 12-201
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Lipid Metabolism Disorder
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — Magnetic Resonance Spectroscopy; Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isocaloric diet (7 days) (Placebo Comparator): Protocole A
  Interventions: Dietary Supplement: isocaloric diet; Other: Liquid meal; Radiation: PET imaging; Other: perfusions of stable tracers; Device: Indirect calorimetry
- Hypercaloric diet enriched with carbohydrate food (7 days) (Experimental): Protocole B
  Interventions: Dietary Supplement: Hypercaloric diet; Other: Liquid meal; Radiation: PET imaging; Other: perfusions of stable tracers; Device: Indirect calorimetry

INTERVENTIONS:
Dietary Supplement: isocaloric diet — a 7-day isocaloric diet
  Arms: Isocaloric diet (7 days)
Dietary Supplement: Hypercaloric diet — A 7-day hypercaloric diet supplemented with carbohydrate-rich food (+ 50% of the subject's energy needs).
  Arms: Hypercaloric diet enriched with carbohydrate food (7 days)
Other: Liquid meal
Radiation: PET imaging
Other: perfusions of stable tracers
Device: Indirect calorimetry

SUMMARY:
The present research protocol will analyze whether a short-term modification (one week) of dietary habits would have an impact on the postprandial metabolism of dietary fatty acids and on their uptake by non-adipose tissues, in healthy subjects.

Each subject will participate in two protocols randomly determined and separated by a period of one month: a 7-day isocaloric diet (Protocol A) and a 7-day carbohydrate-rich diet containing +50% of the subject's energy needs. (Protocol B).

At the end of each diet, the subject will go through a postprandial metabolic study of 8 hours where different parameters will be measured thanks to PET imaging and perfusions of stables isotopes.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects: subjects with normal glucose tolerance determined according to an oral glucose tolerance test and with a BMI above 25 kg/m2 without first degree of familial history of type 2 diabetes (parents, siblings).

Exclusion Criteria:

* overt cardiovascular disease as assessed by medical history, physical exam, and abnormal ECG
* treatment with a fibrate, thiazolidinedione, beta-blocker or other drug known to affect lipid or carbohydrate metabolism (except statins, metformin, and other antihypertensive agents that can be safely interrupted)
* presence of liver or renal disease, uncontrolled thyroid disorder, previous pancreatitis, bleeding disorder, or other major illness
* smoking (>1 cigarette/day) and/or consumption of >2 alcoholic beverages per day
* prior history or current fasting plasma cholesterol level > 7 mmol/l or fasting TG > 5 mmol/l
* any other contraindication to temporarily interrupt current meds for lipids or hypertension
* being pregnant
* not be barren

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
whole-body organ-specific Dietary Fatty Acid (DFA) partitioning | 2 months
  will be determined by whole-body CT (16 mA) followed by PET acquisition of 18FTHA
Left ventricular function by Positron Emiting Positron (PET) ventriculography | 2 months
  will be determined using 11C-acetate PET/CT. 180 MBq will be administered by bolus injection at fasting. After a transmission scan and regional CT (40mA), a 30-min dynamic list-mode PET acquisition will be performed on a 18 cm-high thoraco-abdominal segment to include the left cardiac ventricle and most of the liver on a Philips Gemini TOF PET/CT

SECONDARY OUTCOMES:
Cardiac DFA uptake | 2 months
  will be assessed using PET/CT method with oral administration of 18FTHA followed by a 30 min. dynamic PET acquisition
Cardiac and hepatic oxidative metabolism index | 2 months
  will be determined using 11C-acetate PET/CT followed by a 30 minutes dynamic PET acquisition.
Cardiac and hepatic blood flow | 2 months
  will be determined using 11C-acetate PET/CT followed by a 30 minutes dynamic PET acquisition..
metabolites appearance rate | 6 months
  will be determined by perfusion of stable isotope tracers
energy metabolism (whole body production) | 4 months
  by indirect calorimetry
hormonal responses | 4 months
  analysed by colorimetric and Elisa tests
Insulin sensitivity | 4 months
  will be determined using the HOMA-IR (based on fasting insulin and glucose) levels
Insulin secretion rate | 4 months
  will be assessed using deconvolution of plasma C-peptide with standard Cpeptide kinetic parameters
β-cell function | 4 months
  will be assessed by calculation of the disposition index (DI) that is insulin secretion in response to the ambient insulin
Anthropometric parameters | 2 months
  will be measured at each postprandial metabolic study

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Montastier E, Ye RZ, Noll C, Bouffard L, Fortin M, Frisch F, Phoenix S, Guerin B, Turcotte EE, Lewis GF, Carpentier AC. Increased postprandial nonesterified fatty acid efflux from adipose tissue in prediabetes is offset by enhanced dietary fatty acid adipose trapping. Am J Physiol Endocrinol Metab. 2021 Jun 1;320(6):E1093-E1106. doi: 10.1152/ajpendo.00619.2020. Epub 2021 Apr 19. PMID 33870714